CLINICAL TRIAL: NCT00322205
Title: Bio-behavioral Lung Cancer Prevention Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health (NIH) (NIH)
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 703463; NCT00326755 (obsolete NCT alias)
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2006-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion

INTERVENTIONS:
Drug: zyban

SUMMARY:
The overall goal of this research is to increase our understanding of the role of individual genetic differences in response to bupropion treatment and the psychobiological mechanisms by which genetic and treatment factors interact in the smoking cessation process. The ultimate objective is to provide information necessary to match bupropion vs. behavioral counseling cessation treatment to those smokers with the greatest need and likelihood of benefit. This study is a double-blind randomized placebo-controlled clinical trial of bupropion HCL (brand name Zyban) in adult male and female smokers. The factorial design includes one treatment factor (bupropion 300 mg/day + counseling vs. placebo + counseling) and several subject factors (e.g. genotype, personality). Smoking history, psychological status will be assessed at baseline and blood will be drawn for genotyping. Bupropion or placebo will be delivered over a 10-week treatment period and subjects will be instructed to quit smoking after two weeks of medication (week 3 of treatment). All subjects will also receive a 7-week group behavioral smoking cessation treatment (over an 11 week period). This study may yield information that will help clinicians identify the most effective smoking cessation treatment for a particular patient, based on his/her background.

ELIGIBILITY:
Inclusion Criteria:

Eligible smokers will be those currently smoking at least 10 cigarettes a day.

Exclusion Criteria:

Exclusionary criteria are: planning a pregnancy, pregnancy, lactating, seizure disorder, history of head trauma or prior seizure, family history of a seizure disorder, brain (or CNS) tumor, history of or currently diagnosed with bulimia or anorexia nervosa, diabetes treated with oral hypoglycemics or insulin, excessive use of alcohol or alcoholism, current addiction to opiates, cocaine, or stimulants, use of other drugs containing bupropion (e.g., Wellbutrin, Wellbutrin SR), allergy to bupropion, currently taking particular medications (e.g., monoamine oxidase inhibitor, antipsychotics, antidepressants, theophylline, systemic steroids, over-the-counter stimulants and anorectics), recently taken a MAOI (less than 14 days) or a recent discontinuation of a benzodiazepine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 555
Dates: Start 1999-06; Study Completion 2002-03

PRIMARY OUTCOMES:
Continuous abstinence: measured at end of treatment and at 6- and 12- months after cessation.

SECONDARY OUTCOMES:
Short-term quit rates using 7-day and 30-day point prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Principal Investigator — University of Pennsylvania
Locations (1):
- State University of New York, Buffalo, New York, United States

REFERENCES:
- [Result] Lerman C, Jepson C, Wileyto EP, Epstein LH, Rukstalis M, Patterson F, Kaufmann V, Restine S, Hawk L, Niaura R, Berrettini W. Role of functional genetic variation in the dopamine D2 receptor (DRD2) in response to bupropion and nicotine replacement therapy for tobacco dependence: results of two randomized clinical trials. Neuropsychopharmacology. 2006 Jan;31(1):231-42. doi: 10.1038/sj.npp.1300861. PMID 16123753
- [Result] Wileyto EP, Patterson F, Niaura R, Epstein LH, Brown RA, Audrain-McGovern J, Hawk LW Jr, Lerman C. Recurrent event analysis of lapse and recovery in a smoking cessation clinical trial using bupropion. Nicotine Tob Res. 2005 Apr;7(2):257-68. doi: 10.1080/14622200500055673. PMID 16036283
- [Result] Lerman C, Niaura R, Collins BN, Wileyto P, Audrain-McGovern J, Pinto A, Hawk L, Epstein LH. Effect of bupropion on depression symptoms in a smoking cessation clinical trial. Psychol Addict Behav. 2004 Dec;18(4):362-6. doi: 10.1037/0893-164X.18.4.362. PMID 15631608
- [Result] Wileyto P, Patterson F, Niaura R, Epstein L, Brown R, Audrain-McGovern J, Hawk L, Lerman C, Patterson F. Do small lapses predict relapse to smoking behavior under bupropion treatment? Nicotine Tob Res. 2004 Apr;6(2):357-66. doi: 10.1080/1462220042000202463. PMID 15203809
- [Result] Lerman C, Berrettini W, Pinto A, Patterson F, Crystal-Mansour S, Wileyto EP, Restine SL, Leonard DG, Shields PG, Epstein LH. Changes in food reward following smoking cessation: a pharmacogenetic investigation. Psychopharmacology (Berl). 2004 Aug;174(4):571-7. doi: 10.1007/s00213-004-1823-9. Epub 2004 Apr 27. PMID 15138759
- [Result] Collins BN, Wileyto EP, Patterson F, Rukstalis M, Audrain-McGovern J, Kaufmann V, Pinto A, Hawk L, Niaura R, Epstein LH, Lerman C. Gender differences in smoking cessation in a placebo-controlled trial of bupropion with behavioral counseling. Nicotine Tob Res. 2004 Feb;6(1):27-37. doi: 10.1080/14622200310001656830. PMID 14982685
- [Result] Lerman C, Shields PG, Wileyto EP, Audrain J, Pinto A, Hawk L, Krishnan S, Niaura R, Epstein L. Pharmacogenetic investigation of smoking cessation treatment. Pharmacogenetics. 2002 Nov;12(8):627-34. doi: 10.1097/00008571-200211000-00007. PMID 12439223
- [Result] Lerman C, Roth D, Kaufmann V, Audrain J, Hawk L, Liu A, Niaura R, Epstein L. Mediating mechanisms for the impact of bupropion in smoking cessation treatment. Drug Alcohol Depend. 2002 Jul 1;67(2):219-23. doi: 10.1016/s0376-8716(02)00067-4. PMID 12095672
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Ashare RL, Wileyto EP, Perkins KA, Schnoll RA. The first 7 days of a quit attempt predicts relapse: validation of a measure for screening medications for nicotine dependence. J Addict Med. 2013 Jul-Aug;7(4):249-54. doi: 10.1097/ADM.0b013e31829363e1. PMID 23669629
- [Derived] Javitz HS, Lerman C, Swan GE. Comparative dynamics of four smoking withdrawal symptom scales. Addiction. 2012 Aug;107(8):1501-11. doi: 10.1111/j.1360-0443.2012.03838.x. Epub 2012 Apr 17. PMID 22321019